CLINICAL TRIAL: NCT01629303
Title: Efficacy of Sacral Nerve Modulation in Severe Refractory Constipation
Acronym: CONSTIMOD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHUBX 2011/23
Record Dates: First submitted 2012-06-11; First posted 2012-06-27 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Constipation
Keywords: constipation; sacral nerve modulation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm on-off (Experimental): After the definitive implantation, stimulators are placed in position OFF during 8 weeks.
  Then all the stimulators are switched OFF for 15 days. Finally stimulators are switched ON for the second arm during 8 weeks
  Interventions: Procedure: sacral nerve modulation
- Arm off-on (Experimental): After the definitive implantation, stimulators are placed in position ON during 8 weeks.
  Then all the stimulators are switched OFF for 15 days. Finally stimulators are maintained in position OFF during 8 weeks
  Interventions: Procedure: sacral nerve modulation

INTERVENTIONS:
Procedure: sacral nerve modulation — After the definitive implantation, stimulators are placed in position ON (arm on-off) or OFF (arm off-on) for the first arm and in position OFF for the second arm during 8 weeks.
  Then all the stimulators are switched OFF (both first and second arms) for 15 days.
  Finally stimulators are maintained in position OFF for the first arm and switched ON for the second arm during 8 weeks

SUMMARY:
Subjects with refractory chronic constipation are offered two conventional therapeutic strategies: either medical treatment, either surgery (in the case of medication failure). Nevertheless, a procedure less invasive than surgery could be an alternative strategy: the sacral nerve modulation. This procedure consists in stimulating the nerves which control the contractions of the colon and so the defecation phenomenon. Several open trials have suggested that sacral nerve modulation may be effective in reducing constipation and related symptoms. The aim of this randomized clinical trial is to assess the efficacy of the sacral nerve stimulation in patients with constipation.

DETAILED DESCRIPTION:
The prevalence of constipation is 2-27% in Western countries. For patients failing medical treatment (laxatives, biofeedback), a surgical solution may be considered (subtotal colectomy). But results are variable and it puts them at risk of functional sequelae.

Sacral nerve modulation is a minimally invasive procedure compared with the standard surgical support (colectomy) and reversible, which consists in two stages. First, a 3-week temporary stimulation test allows verifying the efficacy of neuromodulation. If the test is positive, the stimulating electrode is definitely implanted. Risks related to the procedure (infection, pain) are much smaller than those associated with a conventional surgical support.

Non comparative studies conducted with 19 and 62 patients showed that 40-73% of implanted patients have an improvement of their constipation and could benefit of permanent implantation with good results in medium term.

The primary objective of the investigators study is to evaluate the short-term efficacy (percentage of responders at 2 months) of sacral nerve modulation in the treatment of severe chronic constipation.

This is a cross-over designed, double-blinded, French multicenter clinical trial, including two periods: 2 months of stimulation ON and 2 months of stimulation OFF. Between these two periods, a 15-days period of "wash-out" will be respected during which all patients will be in OFF mode (4.5 months in total). This period of 4.5 months will be extended by a follow-up period of 7 months during which all patients will be treated (stimulation ON).

If this trial showed efficiency of this procedure, patients with severe refractory constipation could benefit of a sacral nerve modulation test before considering a surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Constipation defined by at least two of the following criteria :

  * Frequency of 2 stools or less per week
  * Severe outlet constipation, i.e. need to use digital extraction or enemas more than 25% of time
  * Sensation of incomplete evacuation more than 25% of time
* Refractory constipation since at least 1 year to medical treatment (drug treatment and/or biofeedback) conducted in the centre (failure or intolerance to laxative osmotic treatments, stimulants, and prucalopride) for which surgery is discussed
* Patients supported in the centre for at least 3 months before inclusion
* Patients having social security system
* Patients having read and signed informed consent form

Exclusion Criteria:

* Constipation secondary to ano-rectal malformation, surgical sequel, colorectal or anal organic lesions, or pelvi-perineal static disorder indicated for surgical treatment
* Constipation secondary to neurological pathology and/or concomitant treatments intake (opiates, anticholinergic agents)
* Partial colectomy history
* Patients in whom implantation of stimulating electrode is impossible due to anatomical reasons (e.g. sacral agenesis)
* Pregnant female patients or with childbearing potential without adequate contraceptive barrier (oestrogen-progesterone contraceptives or intra-uterine device)
* Skin disease associated with a risk of infection - in the opinion of the investigator
* Patient with pacemaker or defibrillator
* Patient exposed to resonance magnetic imaging
* Psychiatric disease incompatible with use of the treatment - in the opinion of the investigator
* Patient misunderstanding oral and written French language
* Patient participating to another study
* Patients who don't complete the first diary without missing data (concerning items used to define the primary endpoint)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-06; Primary Completion 2013-11 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Percentage of patients showing a positive response to sacral nerve stimulation at 2 months | 2 months of the stimualtion period
  Percentage of patients showing a positive response to sacral nerve stimulation during the period " ON " compared with the period " OFF " based on an objective assessment of the number of feces and their characteristics

SECONDARY OUTCOMES:
Clinical characteristics, manometry data, Wexner score of responders to stimulation during the temporary stimulation test (period before the permanent implantation) | 3 weeks between temporary and permanent implantations
Clinical characteristics, manometry data, Wexner score of responders to short-term stimulation | 2 months after permanent implantation
Efficacy of neuromodulation | 1 year after permanent implantation
  Efficacy of neuromodulation (percentage of positive responders) at 1 year
Manometry data, Wexner, QoL and EVA scores, time of colonic transit of responders to prolonged stimulation | 1 year after permanent implantation
To evaluate the investigator opinion about the neuromodulation response, using the patient diary. | 1 year after permanent implantation

CONTACTS AND LOCATIONS:
Overall Officials: Frank ZERBIB, Professor, Principal Investigator — University Hospital, Bordeaux; Genevieve CHENE, Professor, Study Chair — University Hospital, Bordeaux
Locations (11):
- France (11):
  - Service d'hépato-gastroentérologie et oncologie digestive, Bordeaux, Bordeaux
  - Service d' Hépato-gastro-entérologie, CHU de Limoges, Limoges
  - Service d'exploration fonctionnelle digestive -Hospices Civils de Lyon, Lyon, Lyon
  - : Clinique de chirurgie digestive et endocrinienne. Institut des Maladies de l'Appareil Digestif (IMAD, Nantes, Nantes
  - Service d'hépato-gastroentérologie - CHU estaing, Clermont-Ferrand
  - Service de gastroentérologie - AP HP, Colombes
  - Service de Chirurgie générale - CHU de Grenoble, Grenoble
  - Service de gastroentérologie - hopital nord -AP-HM, Marseille
  - SMAD CHU Pontchaillou -Rennes, Rennes
  - Service de physiologie digestive, urinaire, respiratoire et sportive - CHU de rouen, Rouen
  - Service d'hépato-gastroentérologie et explorations fonctionnelles digestives - CHU de Tours, Tours

REFERENCES:
- [Derived] Zerbib F, Siproudhis L, Lehur PA, Germain C, Mion F, Leroi AM, Coffin B, Le Sidaner A, Vitton V, Bouyssou-Cellier C, Chene G; CONSTIMOD study investigators. Randomized clinical trial of sacral nerve stimulation for refractory constipation. Br J Surg. 2017 Feb;104(3):205-213. doi: 10.1002/bjs.10326. Epub 2016 Oct 25. PMID 27779312